CLINICAL TRIAL: NCT06614205
Title: Tumor Absorbed Dose-Response Relationship in Patients Treated With 177Lu-DOTATATE for Meningioma
Acronym: DATUM
Status: Completed | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, BOURSIER Caroline, Principal Investigator, Central Hospital, Nancy, France
Other Study IDs: 2024PI102
Record Dates: First submitted 2024-06-06; First posted 2024-09-26 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-02

CONDITIONS: Meningioma of Brain
Keywords: meningioma; theragnostic; dosimetry
MeSH Terms: conditions — Meningioma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients treated with 177Lu-DOTATATE for meningioma: Patients treated with 177Lu-DOTATATE for meningioma at the Nancy's hospital who met the treatment criteria of the Compassionate Prescribing Framework and received a scintigraphy at D1, D4 and D7 (± 1 day)
  Interventions: Diagnostic Test: tumoral dosimetry by scintigraphy

INTERVENTIONS:
Diagnostic Test: tumoral dosimetry by scintigraphy — The tumoral dosimetry has been done on patient after treatment by 177Lu-DOTATATE Theses patients performed a scintigraphy exam at D1, D4 and D7 after the treatment

SUMMARY:
The hypothesis for this study is that there is a dose-response relationship in patients treated with 177Lu-DOTATATE for meningiomas.

DETAILED DESCRIPTION:
Dosimetry is essential for Peptide Receptor Radionuclide Therapy (PRRT) of meningiomas, to predict efficacy and dose-effect relationships at the individual level, and to move towards personalized medicine. Due to the increasing therapeutic applications of Lutathera, the European Association of Nuclear Medicine (EANM) recently issued recommendations on the dosimetry of 177Lu-labeled somatostatin analogues. Nevertheless, despite these recommendations, the evaluation of meningioma tumor dosimetry in Peptide Receptor Radionuclide Therapy studies is not systematic, which has not enabled us to clearly determine the dose delivered to the meningioma lesion in these treatments and the possible dose-response relationship in this type of treatment.

ELIGIBILITY:
Inclusion Criteria:

* patients treated for menigioma at nancy hospital
* patients who performed 3 scintigraphics exams during there treatment

Exclusion Criteria:

* patients deprived of liberty
* patient who refused to collect data retrospectively

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patients treated with 177Lu-DOTATATE for meningioma at Nancy University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-02-25 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracy for progression free survival | Day 1
  Accuracy of tumor dosimetry to predict 6-month progression-free survival.

SECONDARY OUTCOMES:
Diagnostic accuracy for overal survival | Day 1
  Accuracy of tumoral dosimetry in predicting 6-month overall survival

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - CHRU de NANCY, Vandœuvre-lès-Nancy
  - Nuclear medicine Department CHRU de NANCY, Vandœuvre-lès-Nancy

IPD SHARING:
Plan to Share IPD: No